CLINICAL TRIAL: NCT03492944
Title: Contrast-Enhanced Ultrasound Evaluation of Bowel Wall Inflammation in Pediatric Crohn's Disease: Comparison to CT and MRI Enterography
Brief Title: Contrast Enhanced Ultrasound in Human Crohn's Disease-Lumason
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN_Lumason Crohns_001
Record Dates: First submitted 2018-02-12; First posted 2018-04-10 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Ultrasound Microbubble Contrast Agent: All subjects will receive intravenous Lumason microbubble contrast agent; there is no comparative ultrasound contrast agent. Contrast Enhanced Ultrasound findings/results will be correlated with comparable, clinically performed, CTE/MRE findings/results
  Interventions: Drug: Ultrasound Microbubble Contrast Agent; Device: Ultrasound Imaging

INTERVENTIONS:
Drug: Ultrasound Microbubble Contrast Agent — Patients undergoing a clinically ordered CT or MRI Enterography for Crohn disease will be recruited to undergo a contrast enhanced ultrasound study of the bowel
  Other Names: Lumason
Device: Ultrasound Imaging — Patients undergoing a clinically ordered CT or MRI Enterography for Crohn disease will be recruited to undergo a contrast enhanced ultrasound study of the bowel

SUMMARY:
The investigators plan to compare contrast-enhanced ultrasound to CT and MRI for the detection and quantification of intestinal inflammation in the the setting of pediatric small bowel Crohns disease

DETAILED DESCRIPTION:
The proposed study will investigate the use of an FDA-approved ultrasound microbubble contrast agent (Lumason; Bracco Diagnostics) in pediatric and adult Crohn's disease patients undergoing either MR enterography (MRE, or MRI of the bowel) or CT enterography (CTE, or CT of the bowel). In April 2016, Lumason was FDA approved for intravenous administration and imaging of the liver in children. Imaging of the bowel will employ an identical administration method to that described for liver imaging, but the ultrasound transducer will be placed over the affected intestines as opposed to liver.

ELIGIBILITY:
Inclusion Criteria:

* histologic evidence of small bowel Crohn's disease, or clinical evidence of disease (including radiologic confirmation [either CT or MRI] and receiving medical therapy for Crohn's disease).
* Between ages 10 and 18 years.
* Undergoing clinically-indicated CTE or MRE with evidence of active disease based on pediatric gastroenterologist clinical assessment

Exclusion Criteria:

* Patients under the age of 10 or over the age of 18.
* Pregnancy or breast feeding. Urine pregnancy testing will be performed on all female study participants of reproductive potential.
* Obesity/body habitus preventing visualization of small bowel affected by Crohn's disease by ultrasound (Body mass index ≥30 kg/m2
* Subject inability/unwillingness to consent or child assent, including severe developmental delay/mental retardation.
* Prior allergic-like reaction or other severe adverse event to Lumason or any of the active ingredients in Lumason (SPECIFIC CONTRAINDICATION from Package Insert).
* Known unstable cardiopulmonary conditions (including any history of acute myocardial infarction/acute coronary artery syndrome, arrhythmia, and congestive heart failure), ongoing acute or chronic kidney disease (eGFR <30 ml/min), moderate/severe chronic lung disease, and end-stage liver disease.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We plan to recruit approximately 25 subjects, 10-18 years of age, with known small bowel Crohn disease undergoing clinically indicated Computed Tomography Enterography (CTE) or Magnetic Resonance Enterography (MRE)imaging
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Degree of bowel wall enhancement | 2 years
  Percent hyperenhancement (compared to normal bowel loops)

SECONDARY OUTCOMES:
Overall Disease Status for imaged section | 2 years
  status of inactive, mild activity, moderate activity and severe activity
Degree of mesenteric inflammation | 2 years
  Inflammation assessed as none, mild, moderate, severe
Maximum Bowel Wall Thickness | 2 years
  Measured

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dillman, MD,MSc, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Research data including identifying information about participants will only be accessible to CCHMC study personnel. De-identified data including images will be shared with scientists at Bracco Diagnostics. No identifiable data will be shared

REFERENCES:
- [Background] Adler J, Punglia DR, Dillman JR, Polydorides AD, Dave M, Al-Hawary MM, Platt JF, McKenna BJ, Zimmermann EM. Computed tomography enterography findings correlate with tissue inflammation, not fibrosis in resected small bowel Crohn's disease. Inflamm Bowel Dis. 2012 May;18(5):849-56. doi: 10.1002/ibd.21801. Epub 2011 Jun 24. PMID 21710535
- [Background] Girlich C, Jung EM, Huber E, Ott C, Iesalnieks I, Schreyer A, Schacherer D. Comparison between preoperative quantitative assessment of bowel wall vascularization by contrast-enhanced ultrasound and operative macroscopic findings and results of histopathological scoring in Crohn's disease. Ultraschall Med. 2011 Apr;32(2):154-9. doi: 10.1055/s-0029-1245398. Epub 2010 May 6. PMID 20449794
- [Background] Quaia E, Migaleddu V, Baratella E, Pizzolato R, Rossi A, Grotto M, Cova MA. The diagnostic value of small bowel wall vascularity after sulfur hexafluoride-filled microbubble injection in patients with Crohn's disease. Correlation with the therapeutic effectiveness of specific anti-inflammatory treatment. Eur J Radiol. 2009 Mar;69(3):438-44. doi: 10.1016/j.ejrad.2008.10.029. Epub 2008 Dec 12. PMID 19070446
- [Background] Wong DD, Forbes GM, Zelesco M, Mason R, Pawlik J, Mendelson RM. Crohn's disease activity: quantitative contrast-enhanced ultrasound assessment. Abdom Imaging. 2012 Jun;37(3):369-76. doi: 10.1007/s00261-011-9792-z. PMID 21830051
- [Background] De Franco A, Di Veronica A, Armuzzi A, Roberto I, Marzo M, De Pascalis B, De Vitis I, Papa A, Bock E, Danza FM, Bonomo L, Guidi L. Ileal Crohn disease: mural microvascularity quantified with contrast-enhanced US correlates with disease activity. Radiology. 2012 Feb;262(2):680-8. doi: 10.1148/radiol.11110440. Epub 2011 Dec 12. PMID 22157203
- [Background] Girlich C, Schacherer D, Jung EM, Schreyer A, Buttner R. Comparison between a clinical activity index (Harvey-Bradshaw-Index), laboratory inflammation markers and quantitative assessment of bowel wall vascularization by contrast-enhanced ultrasound in Crohn's disease. Eur J Radiol. 2012 Jun;81(6):1105-9. doi: 10.1016/j.ejrad.2011.02.054. Epub 2011 Mar 24. PMID 21439749
- [Background] Ripolles T, Martinez MJ, Paredes JM, Blanc E, Flors L, Delgado F. Crohn disease: correlation of findings at contrast-enhanced US with severity at endoscopy. Radiology. 2009 Oct;253(1):241-8. doi: 10.1148/radiol.2531082269. Epub 2009 Jul 27. PMID 19635834
- [Background] Malago R, D'Onofrio M, Mantovani W, D'Alpaos G, Foti G, Pezzato A, Caliari G, Cusumano D, Benini L, Pozzi Mucelli R. Contrast-enhanced ultrasonography (CEUS) vs. MRI of the small bowel in the evaluation of Crohn's disease activity. Radiol Med. 2012 Mar;117(2):268-81. doi: 10.1007/s11547-011-0783-5. Epub 2012 Jan 21. PMID 22271005
- [Background] Quaia E, De Paoli L, Stocca T, Cabibbo B, Casagrande F, Cova MA. The value of small bowel wall contrast enhancement after sulfur hexafluoride-filled microbubble injection to differentiate inflammatory from fibrotic strictures in patients with Crohn's disease. Ultrasound Med Biol. 2012 Aug;38(8):1324-32. doi: 10.1016/j.ultrasmedbio.2012.04.008. Epub 2012 Jun 13. PMID 22698508
- [Background] Schirin-Sokhan R, Winograd R, Tischendorf S, Wasmuth HE, Streetz K, Tacke F, Trautwein C, Tischendorf JJ. Assessment of inflammatory and fibrotic stenoses in patients with Crohn's disease using contrast-enhanced ultrasound and computerized algorithm: a pilot study. Digestion. 2011;83(4):263-8. doi: 10.1159/000321389. Epub 2011 Jan 28. PMID 21273775
- [Background] Riccabona M, Avni FE, Damasio MB, Ording-Muller LS, Blickman JG, Darge K, Lobo ML, Papadopoulou F, Vivier PH, Willi U. ESPR Uroradiology Task Force and ESUR Paediatric Working Group--Imaging recommendations in paediatric uroradiology, part V: childhood cystic kidney disease, childhood renal transplantation and contrast-enhanced ultrasonography in children. Pediatr Radiol. 2012 Oct;42(10):1275-83. doi: 10.1007/s00247-012-2436-9. Epub 2012 Sep 22. PMID 23001574
- [Background] Main ML, Ryan AC, Davis TE, Albano MP, Kusnetzky LL, Hibberd M. Acute mortality in hospitalized patients undergoing echocardiography with and without an ultrasound contrast agent (multicenter registry results in 4,300,966 consecutive patients). Am J Cardiol. 2008 Dec 15;102(12):1742-6. doi: 10.1016/j.amjcard.2008.08.019. Epub 2008 Oct 23. PMID 19064035
- [Background] McCarville MB, Kaste SC, Hoffer FA, Khan RB, Walton RC, Alpert BS, Furman WL, Li C, Xiong X. Contrast-enhanced sonography of malignant pediatric abdominal and pelvic solid tumors: preliminary safety and feasibility data. Pediatr Radiol. 2012 Jul;42(7):824-33. doi: 10.1007/s00247-011-2338-2. Epub 2012 Jan 17. PMID 22249601
- [Background] Dillman JR, Strouse PJ, Ellis JH, Cohan RH, Jan SC. Incidence and severity of acute allergic-like reactions to i.v. nonionic iodinated contrast material in children. AJR Am J Roentgenol. 2007 Jun;188(6):1643-7. doi: 10.2214/AJR.06.1328. PMID 17515388
- [Background] Wang CL, Cohan RH, Ellis JH, Adusumilli S, Dunnick NR. Frequency, management, and outcome of extravasation of nonionic iodinated contrast medium in 69,657 intravenous injections. Radiology. 2007 Apr;243(1):80-7. doi: 10.1148/radiol.2431060554. PMID 17392249